CLINICAL TRIAL: NCT02404571
Title: The Efficacy and Toxicity of GDP Chemotherapy in Patients With Peripheral T-cell Lymphoma: An Open-label, Single-arm, Phase II Clinical Trial
Brief Title: GDP in Frontline Chemotherapy for Patients With PTCL-NOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mei Dong, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GiFT
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GDP chemotherapy (Experimental): GDP chemotherapy: gemcitabine (1000mg/m2 intravenously over 30 minutes on days 1 and 8), cisplatin (25mg/m2 intravenously over 60 minutes on days 1-3), and dexamethasone (20mg/d orally on days 1-4 and days 11-14), which was administered every 21 days.
  Interventions: Drug: GDP chemotherapy

INTERVENTIONS:
Drug: GDP chemotherapy — gemcitabine (1000mg/m2 intravenously over 30 minutes on days 1 and 8), cisplatin (25mg/m2 intravenously over 60 minutes on days 1-3), and dexamethasone (20mg/d orally on days 1-4 and days 11-14), which was administered every 21 days.

SUMMARY:
This study is to evaluate the efficacy and safety of GDP (gemcitabine, dexamethasone, and cisplatin) chemotherapy in patients with peripheral T-cell lymphoma-NOS as frontline treatment.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas,not otherwise specified constitutes 25.9% of Peripheral T-cell lymphomas and over 15% of all lymphomas by the World Health Organization classification. Because of the rare presentation and evident heterogeneity of PTCL-NOS, optimal frontline therapy for this disease in the modern era remains unclear. Patients have traditionally been treated with anthracycline-containing chemotherapy such as CHOP or CHOP-like regimen used in B-cell NHLs. This strategy is associated with an overall response rate higher than 60%, but the 5-year PFS and OS rates have been reported to be as low as approximately 20-30%.Better therapeutic regimens are in highly need to improve the survival outcome of these patients. The investigators' previous study reported an ORR of 64% in relapsed/refractory PTCL-NOS patients. Therefore, the investigators design this study to evaluate the efficacy and safety of GDP chemotherapy as frontline treatment in patients with PTCL-NOS.

ELIGIBILITY:
Inclusion Criteria:

1. histological and imaging diagnosis of PTCL-NOS based on immunophenotypic and morphologic criteria according to the 2008 World Health Organization classification of lymphomas;
2. newly-diagnosed patients with no prior systemic chemotherapy or stem-cell transplantation treatment.
3. age ≥ 18 years;
4. life expectancy of more 3 months;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
6. at least one measurable lesion;
7. adequate hematologic, hepatic, and renal functions: absolute neutrophil count ≥ 1.5×109/l, platelet count ≥ 100×109/l, total bilirubin ≤ 1.5 × upper limit of normal, AST and ALT ≤ 2 × upper limit of normal, and creatinine ≤ 1.5 mg/dl;
8. informed consent.

Exclusion Criteria:

1. patients who received prior treatment;
2. pregnant or breastfeeding women and women of childbearing potential not employing adequate contraception;
3. patients with second primary cancer (except, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years)
4. patients with defect of central nervous system (CNS) or any psychiatric disorders and CNS metastases
5. other serious illness or medical conditions A. Clinically significant cardiac disease (uncontrolled congestive heart disease despite treatment [NYHA class III or IV], symptomatic coronary artery disease, unstable angina or myocardial infarction, conduction abnormality like grade 2 AV block, serious arrhythmia needed for medication, uncontrolled hypertension) within 6 months prior to study entry B. Liver cirrhosis (≥ Child-Pugh class B) C. History of significant neurologic or psychiatric disorders including dementia or seizures D. Active uncontrolled infection E. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 4-6 cycles

SECONDARY OUTCOMES:
2-year progression-free survival | 2 year
2-year overall survival | 2 year
number of patients with adverse events | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Mei Dong, Principal Investigator — Cancer Hospital and Institute, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC)
Locations (1):
- Cancer Hospital and Institute, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China